CLINICAL TRIAL: NCT00231296
Title: A Clinical Study to Evaluate the Safety and Efficacy of the CryoCor(TM)Cardiac Cryoablation System for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Safety and Efficacy of CryoCor™ Cryoablation for PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-AF-02
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
Keywords: cryoablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment with CryoCor Cryoablation System (Active Comparator): Intervention includes ablation therapy with the CryoCor catheter for the treatment of symptomatic PAF.
  Interventions: Device: Cardiac CryoCor Cryoablation System
- Treatment with standard medical therapy (Active Comparator): Intervention includes treatment with ant-arrhythmic medications alone.
  Interventions: Drug: Medical management

INTERVENTIONS:
Device: Cardiac CryoCor Cryoablation System — Treatment with CryoCor Cardiac Cryoablation system
  Other Names: Ablation with the CryoCor ablation catheter
  Arms: Treatment with CryoCor Cryoablation System
Drug: Medical management — Medical management- treatment with standard medical therapy, which includes anti-arrhythmic medications
  Other Names: AAD treatment
  Arms: Treatment with standard medical therapy

SUMMARY:
A multi-center, randomized, controlled study of cryoablation vs medical management for the treatment of PAF

DETAILED DESCRIPTION:
The purpose of this prospective, randomized multi-center clinical study is to establish the benefits of the CryoCor(TM) Cardiac Cryoablation System for treating symptomatic paroxysmal atrial fibrillation (PAF) in comparison to treatment with anti-arrhythmic medications alone. This study also evaluates the safety profile of the CryoCor(TM) Cardiac Cryoablation System when used in this same setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 episodes of PAF within 6 months
* Refractory to at least one drug
* Therapeutic anticoagulation
* Signed informed consent

Exclusion Criteria:

* Persistent AF
* Structural heart disease
* Prior ablation
* Contraindication present

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety profile of intervention | 12 months
Recurrence of PAF | 12 months

SECONDARY OUTCOMES:
Change in QOL as measured by SF-36 Health Survey | 12 months
  Changes compared to baseline will be measured over a period of 12 months
Change in QOL as measured by Symptom Checklist | 12 months
  Changes compared to baseline will be measured over a period of 12 months
Change in QOL as measured by Arrhythmia Severity scale | 12 months
  Changes compared to baseline will be measured over a period of 12 months
Change in luminal PV measurements | 6 months
Time to treatment failure, post resolution period | Post resolution period (12 months follow-up)
  Time to treatment failure, defined as event monitor documented recurrent atrial fibrillation, post resolution period.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Feld, MD, Principal Investigator — University of California, San Diego
Locations (24):
- United States (24):
  - Regional Cardiology Associates, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - UCSF Medical, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Carle Heart Center, Urbana, Illinois
  - Genesis Health, Davenport, Iowa
  - Iowa Heart Center, Des Moines, Iowa
  - Cardiology Associates of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Heart and Vascular Institute, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Austin Heart, PA, Austin, Texas
  - Methodist Debakey Heart Center, Houston, Texas
  - Tacoma General, Tacoma, Washington
  - Heart Care Associates, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No